CLINICAL TRIAL: NCT05685719
Title: A Study to Evaluate the Relative Bioavailability of Different Strengths of STI-1558 Capsules and the Effect of Strong CYP3A4 Inhibitor (Itraconazole) and Inducer (Rifampin) on the Pharmacokinetics of STI-1558 in Healthy Volunteers
Brief Title: A Study to Evaluate the Relative Bioavailability of STI-1558 and the Effect of Itraconazole and Rifampin on the Pharmacokinetics of STI-1558
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang ACEA Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: MPR-COV-102CN
Record Dates: First submitted 2022-12-21; First posted 2023-01-17 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: COVID-19 Pneumonia
MeSH Terms: interventions — STI-1558; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1: TR (Experimental): Subjects will take a single dose of test product 200mg/capsule on Day 1 of the study, then reference product 100mg/capsule on Day 8 of the study.
  Interventions: Drug: STI-1558
- Part 1: RT (Experimental): Subjects will take a single dose of reference product 100mg/capsule on Day 1 of the study, then test product 200mg/capsule on Day 8 of the study.
  Interventions: Drug: STI-1558
- Part 1: Group 1 (Experimental): Subjects will take a single dose of STI-1558 200mg/capsule on Day 1. Starting from Day 4, subjects will orally take 200mg of itraconazole, q.d, for 6 consecutive days (Day 4 to Day 9). The 5th dose (Day 8) of itraconazole will be co-administered with STI-1558 (200 mg/capsule × 3 capsules) to subjects.
  Interventions: Drug: STI-1558; Drug: Itraconazole
- Part 1: Group 2 (Experimental): Subjects will take a single dose of STI-1558 200mg/capsule on Day 1. Starting from Day 4, subjects will orally take 600mg of rifampin, q.d, for 9 consecutive days (Day 4 to Day 12). The 8th dose (Day 11) of rifampin will be co-administered with STI-1558 (200 mg/capsule × 3 capsules) to subjects.
  Interventions: Drug: STI-1558; Drug: Rifampin

INTERVENTIONS:
Drug: STI-1558 — An oral small molecule prodrug that effectively inhibits the SARS-CoV-2 main protease (Mpro).
Drug: Itraconazole — A strong CYP3A4 inhibitor
  Arms: Part 1: Group 1
Drug: Rifampin — A strong CYP3A4 inducer
  Arms: Part 1: Group 2

SUMMARY:
This is an open-label study. This study includes 2 parts, in which part 1 is a relative BA study, Part 2 is a DDI study. Part 1 and Part 2 could be performed in parallel.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are fully informed of the study and are willing to participate in the study and sign the informed consent document prior to any procedure.
2. Healthy male and female subjects, aged 18 to 45 years (both inclusive).
3. Body mass index (BMI) is between 19 and 24 kg/m2 (both inclusive), and body weight of female subjects ≥ 45 kg, body weight of male subjects ≥ 50 kg.
4. Health status is good, the medical history, vital signs, physical examination, 12- lead ECG, laboratory tests (hematology, blood glucose, blood biochemistry, urinalysis, coagulation test), thyroid function (TSH, FT3, FT4) and serum virology test results are normal or abnormal with no clinical significance (NCS) during the screening period.
5. Female subjects of child-bearing potential must agree to use highly effective contraceptive methods from the screening period to 30 days after the last dose of the study drug, (See Appendix 2 Contraceptive Methods).
6. Male subjects considered fertile must agree to not plan to father a child, not donate sperm, and take effective contraceptive methods from the screening period to 30 days after the last dose of the study drug, (See Appendix 2 Contraceptive Methods).
7. Subjects who are able to communicate well with PI, as well as understand and adhere to the requirements of this study.

Exclusion Criteria:

1. Difficulties in venous blood collection or history of dizziness when encountering blood or needles.
2. Known or suspected pregnancy, or breastfeeding.
3. Has a clinically relevant intolerance or allergy to drugs, or are known or suspected to have hypersensitivity to any ingredient in the STI-1558.
4. Only for Part 2: Known or suspected hypersensitivity to any ingredient in formulations of itraconazole and/or rifampicin (See the product label for the relevant information).
5. Has received an experimental agent (vaccine, drug, biologic, device, blood product or medication) within 1 month or 5 times half-life (whichever is longer) before the first dose of study drug.
6. Has a history of gastrointestinal (such as duodenal ulcer, alimentary tract hemorrhage, etc.), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs as determined by the Principal Investigator (PI, or designee).
7. Has a medical history of other significant diseases (including but not limited to respiratory, circulatory, digestive, hematological, endocrinological, immunological, dermatological, mental and nervous systems, facial diseases and other related diseases).
8. Has a major surgery within 3 months before the first dose of the study drug or plans to undergo surgery during the study.
9. Has a history of febrile illness within 14 days before the first dose of the study drug.
10. Has values above the 1.5 × upper limits of normal (ULN) at screening or Day -1 for the following laboratory measures: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and/or total bilirubin.
11. QTcF interval is prolonged at screening or Day -1 (male: QTcF interval ≥ 450 ms, female: QTcF interval ≥ 470 ms).
12. Vaccinated within 14 days before the first dose of the study drug or plans to be vaccinated during the study.
13. Use of BCRP substrates within 7 days before the first dose of the study drug (see Appendix 3).
14. Use of CYP3A4 strong inducers or inhibitors, or CYP1A2 strong inducers within 7 days before the first dose of the study drug (see Appendix 3).
15. Any marketed medication (prescription and nonprescription) within 14 days or 5 times the half-life (whichever is longer) before the first dose of study drug. (Excluding oral contraceptives, or topical ointments at the discretion of the PI (or designee)).
16. A known history of drug abuse within 2 years before the screening; or positive drug abuse test on Day -1.
17. Blood donation or blood loss of more than 400 mL within 3 months before the screening (excluding menstrual blood loss of women).
18. Weekly alcohol consumption of more than 14 units of alcohol (1 unit of alcohol = 360 mL of beer or 45 mL of spirit with the alcohol content of 40% or 150 mL of wine) in any week within the past 3 months before screening; or intake of alcohol- containing products within 48 hours before the first dose of the study drug, or cannot abstain from any alcohol product during the study, or positive breath alcohol test on Day -1.
19. Smoking history (≥ 5 cigarettes per day) within 3 months before the screening, or cannot abstain from any tobacco products during the study.
20. Excessive drinking of tea, coffee, or caffeine-containing beverage (at least 8 cups per day, 1 cup=250 mL) within 3 months before screening; intake of rich caffeine- or xanthine-containing food or drinks (e.g., coffee, tea, chocolate, cola drinks) within 48 hours before the first dose of the study drug.
21. Intake of food, juice, or drink containing grapefruit, lime, cinchona peel, or quinine within 48 h before the first dose of the study drug.
22. The results of serum virology test are positive or exceed the upper limit of the reference range, including: hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, human immunodeficiency virus (HIV) antibody, or treponema pallidum antibody (TP-Ab).
23. Subjects who are judged as not eligible to participate in this study by the PI (or designee).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2023-01-04 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-11-03 (Actual)

PRIMARY OUTCOMES:
Comparison of Area Under the Curve (AUC) from time 0 to last time point(AUC0-t) profiles of two different oral strength of STI-1558 to determine the Relative Bioavailability | Up to 2 weeks.
  To compare AUC0-t of a single 600mg dose of two different oral strength of STI-1558（200 mg/capsule × 3 capsules and 100 mg/capsule × 6 capsules）in healthy adult, human subjects under fasting conditions, to establish relative bioavailability.
Comparison of AUC from time 0 extrapolated to infinity(AUC0-inf ) profiles of two different oral strength of STI-1558 to determine the Relative Bioavailability | Up to 2 weeks.
  To compare AUC0-inf of a single 600mg dose of two different oral strength of STI-1558（200 mg/capsule × 3 capsules and 100 mg/capsule × 6 capsules）in healthy adult, human subjects under fasting conditions, to establish relative bioavailability.
Comparison of maximum observed concentration(Cmax) profiles of two different oral strength of STI-1558 to determine the Relative Bioavailability | Up to 2 weeks.
  To compare Cmax of a single 600mg dose of two different oral strength of STI-1558（200 mg/capsule × 3 capsules and 100 mg/capsule × 6 capsules）in healthy adult, human subjects under fasting conditions, to establish relative bioavailability.
To determine the effect of repeat doses of a strong CYP3A4 inhibitor (itraconazole) on the pharmacokinetics(PK) of STI-1558 by collecting serum at protocol-specified time points: Cmax | Up to 3 weeks.
To determine the effect of repeat doses of a strong CYP3A4 inhibitor (itraconazole) on the PK of STI-1558 by collecting serum at protocol-specified time points: AUC0-t | Up to 3 weeks.
To determine the effect of repeat doses of a strong CYP3A4 inhibitor (itraconazole) on the PK of STI-1558 by collecting serum at protocol-specified time points: AUC0-inf. | Up to 3 weeks.
To determine the effect of repeat doses of a strong CYP3A4 inducer (rifampin) on the PK of STI-1558 by collecting serum at protocol-specified time points: Cmax | Up to 3 weeks.
To determine the effect of repeat doses of a strong CYP3A4 inducer (rifampin) on the PK of STI-1558 by collecting serum at protocol-specified time points: AUC0-t | Up to 3 weeks.
To determine the effect of repeat doses of a strong CYP3A4 inducer (rifampin) on the PK of STI-1558 by collecting serum at protocol-specified time points: AUC0-inf | Up to 3 weeks.

SECONDARY OUTCOMES:
Cmax of AC1115(an active metabolite of STI-1558) | Up to 2 weeks for part 1 and 3 weeks for part 2.
AUC0-t of AC1115(an active metabolite of STI-1558) | Up to 2 weeks for part 1 and 3 weeks for part 2.
AUC0-inf of AC1115(an active metabolite of STI-1558) | Up to 2 weeks for part 1 and 3 weeks for part 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No